CLINICAL TRIAL: NCT01162460
Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2-093) as Monotherapy for Patients With Newly Diagnosed Partial-onset Seizures:a Double-blind, Randomized, Active-controlled, Parallel-group, Multicenter Clinical Study
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate as Monotherapy for Patients With Newly Diagnosed Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-311
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbamazepine controlled release (Active Comparator)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Eslicarbazepine acetate (Experimental)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)

INTERVENTIONS:
Drug: Eslicarbazepine acetate (BIA 2-093) — Week 1 and 2 either 400mg/day Eslicarbazepine acetate (ESL) or 200mg/day Carbamazepine controlled release(CBZ-CR); Week 3 onwards either 800mg/day Eslicarbazepine acetate or 400mg/day CBZ-CR; this dose then to be maintained unless a subject has a seizure.
  Subjects experiencing a seizure will have their assigned treatment dose increased to ESL 1200mg/day or CBZ 800mg/day.
  Should a subject have another seizure, their assigned treatment is to be increased to ESL 1600mg/day or CBZ 1200mg/day.
  Subjects who remain seizure free for 26 weeks at any dose in an Evaluation Period will continue to receive the allocated treatment under double-blind conditions.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of eslicarbazepine acetate (BIA 2-093) as monotherapy for patients with newly diagnosed partial-onset seizures.

DETAILED DESCRIPTION:
Epilepsy affects more than 50 million adults and children worldwide. Prevalence estimates in the total population vary from 4 to 8 per 1000 subjects. Anti-epileptic drugs (AEDs) are the major intervention and approximately 60% of newly diagnosed patients are seizure free on a single AED, but about 40% are not satisfactorily controlled and 25% suffer from significant adverse events (AEs). This lack of seizure control and unsatisfactory tolerability means there is still a need for new, effective AEDs that can be used as monotherapy.

Given the efficacy of ESL in controlling partial onset seizures, the good tolerability and the convenience of QD dosing instead of twice daily (BID) dosing, ESL could offer a beneficial alternative as a first-line therapy in patients newly diagnosed with epilepsy experiencing partial-onset seizures. This study aims to demonstrate the efficacy and safety of ESL as a monotherapy treatment for this patient population proving non-inferiority to a standard therapy, Carbamazepine controlled release (CBZ-CR).

ELIGIBILITY:
For inclusion in the study, subjects must fulfill all of the following at the time points indicated:

Visit 1 (Days -1 to -7; Screening)

* Have signed an informed consent before undergoing any study-related activities. Subjects of Asian ancestry (subjects with a direct ancestor of Asian origin, irrespective of the generational difference) are required to give written informed consent for genotyping.
* Male or female ≥18 years of age.
* Newly diagnosed epilepsy with at least 2 well documented, unprovoked, clinically evaluated and classified partial seizures (with or without secondary generalization) with clear focal origin, documented clinically OR by electroencephalogram (EEG) OR by imaging studies, within 12 months of Visit 1. In this context, seizures that occur within a period of 48 hours are counted as one seizure.
* At least 1 seizure during the previous 3 months.
* Demonstrated cooperation and willingness to complete all aspects of the study.
* Female subjects without childbearing potential (2 years postmenopausal, bilateral oophorectomy or tubal ligation, or complete hysterectomy) are eligible. Female subjects with childbearing potential must not be pregnant as confirmed by a negative serum ß-human chorionic gonadotropin (hCG) test and sexually active females must be using a medically acceptable effective non-hormonal method of contraception for the duration of the study and until the Post-study visit (PSV).

Visit A1 (Day 1; Randomization and start of double-blind treatment period)

* Have satisfactorily completed the electronic subject diary (eDiary).
* Female subjects with childbearing potential must not be pregnant as confirmed by a negative urine pregnancy test and sexually active females must be using a medically acceptable effective non-hormonal method of contraception for the duration of the study and until the PSV.

Subjects having any of the following at the time points indicated are to be excluded from the study:

Visit 1 (Days -1 to -7)

* History of pseudo-seizures
* Seizures occurring only in clusters.
* History of absence, myoclonic, clonic, tonic, or atonic seizures.
* Documented EEG within 12 months of Visit 1 suggestive of primarily generalized epilepsy.
* History of status epilepticus within the 3 months prior to Visit 1.
* Known progressive neurologic disorder (progressive brain disease, epilepsy secondary to progressive cerebral lesion) as assessed by magnetic resonance imaging or computer tomography.
* Former or current use of any anti-epileptic drug (AED), except for the use of a single AED for a maximum duration of 2 weeks before Visit 1.
* Previous use of ESL or carbamazepine (CBZ).
* Using mono-amine oxidase inhibitors (MAOIs), tricyclic antidepressants, nefazodone, isoniazid, or protease inhibitors or any other anti-retroviral agents (e.g. efavirez) that may raise the levels of CBZ-CR.
* Known hypersensitivity to carboxamide derivatives or tricyclic antidepressants.
* History of uncontrolled psychiatric illness or mood disorder requiring electro-convulsive or drug therapy within the previous 6 months, a history of suicide attempt, schizophrenia, chronic treatment with benzodiazepines (except short-acting benzodiazepines) or barbiturates.
* Judged clinically to have a suicidal risk in the opinion of the investigator based upon a clinical interview and the Columbia Suicide-Severity Rating Scale (C-SSRS).
* History of alcohol, drug, or medication abuse within the last 2 years.
* Uncontrolled cardiac (including atrioventricular block and other clinically significant electrocardiographic abnormalities), renal, hepatic, endocrine, gastrointestinal, metabolic, hematological, or oncology disorder.
* History of bone marrow depression.
* History of hepatic porphyrias (e.g. acute intermittent porphyria, variegate porphyria, porphyria cutanea tarda).
* Relevant clinical laboratory abnormalities (e.g. sodium <130 mmol/L, alanine or aspartate transaminases >2 x the upper limit of normal, white blood cell count <3000 cells/mm3) (measured at Visit 1).
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (measured at Visit 1).
* Subjects of Asian ancestry who test positive for the presence of the HLA-B*1502 allele.
* Pregnancy or lactating.
* Participation in other drug clinical trial within the last 2 months or having received an investigational medicinal product (IMP) within 5 half-lives of that IMP, whichever is longer.
* Any other condition or circumstance that, in the opinion of the investigator, could compromise the subject's ability to comply with the study protocol.

Visit A1 (Day 1)

* Former or current use of any AED, except for the use of a single AED for a maximum duration of 2 weeks before Visit 1 and with a drug-free period of at least 5 days before Visit A1. Benzodiazepines are allowed, no more than twice a week, for an epileptic indication and as rescue medication during the ≥5-day drug-free period.
* Using prohibited medication.
* Pregnancy.
* Any other condition or circumstance that, in the opinion of the investigator, could compromise the subject's ability to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Actual)
Dates: Start 2010-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the proportion of subjects in the PP set who are seizure free for the entire 26-week Evaluation Period at the last received dose level. | 26 weeks

SECONDARY OUTCOMES:
Proportion of subjects in the ITT set without a seizure during the 26-week Evaluation Period at the last evaluated dose. | 26 weeks
Proportion of subjects without a seizure during the 26-week Evaluation Period at the last evaluated dose. | 26 weeks
Proportion of seizure-free subjects during 1 year of treatment at the last evaluated dose, where the end of the 1-year period is defined as the same start date as for the 26-week evaluation +365 days. | 52 weeks
Time to first seizure at the last evaluated dose set. | up to 183 weeks
QOLIE-31 and Bond-Lader VAS | 26 weeks; up to 183 weeks
  Changes in quality of life assessed using the QOLIE-31 (Overall score, subscores covering emotional well-being, social functioning, energy/fatigue, cognitive functioning, seizure worry, medication effects and assessment of overall health).
Treatment retention time at the last evaluated dose | 26 weeks
  Treatment retention time at the last evaluated dose, where treatment retention time is defined as the time of the first occurrence of one of the following:
  * Withdrawal of IMP due to AEs.
  * Withdrawal of IMP due to lack of efficacy.
Time to treatment failure at the first evaluated dose | 26 weeks
  Time to treatment failure at the first evaluated dose, where time to treatment failure is defined as the time of the first occurrence of 1 of the following:
  * Seizure
  * Withdrawal of IMP due to AEs.
  * Withdrawal of IMP due to lack of efficacy.
seizure freedom | 26 weeks
  Dose level at which subjects reached 26-week seizure freedom.
Adverse Event monitoring | up to 183 weeks
  Incidence of AEs, SAEs, withdrawals, out-of-range laboratory values, abnormal 12-lead ECG and physical examination findings.

CONTACTS AND LOCATIONS:
Locations (1):
- BIAL - Portela & Cª, S.A., S. Mamede Do Coronado, S. Mamede Do Coronado, Portugal